CLINICAL TRIAL: NCT06986629
Title: Effect of Photobiostimulation Versus Pulsed Electromagnetic Field on Quality of Life in Adults With Chronic Rhinosinusitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samar Said Abd Al-Razek Abd Al-Fattah, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Samar-005562
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Photobiostimulation; Pulsed Electromagnetic Filed; Low Level Laser Therapy; Chronic Rhinosinusitis (Diagnosis); Quality of Life
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pulsed electromagnetic therapy (Experimental): This group included twenty adults with chronic rhinosinusitis and received pulsed electromagnetic therapy. This treatment protocol will be carried out three times per week for 8 weeks
  Interventions: Device: pulsed electromagnetic therapy
- Photobiostimulation (Active Comparator): This group included twenty adults with chronic rhinosinusitis and received low level laser therapy. This treatment protocol will be carried out three times per week for 8 weeks
  Interventions: Device: Photobiostimulation
- Self-sinus massage technique (Active Comparator): This group included twenty adults with chronic rhinosinusitis and received the self-sinus massage technique only. This treatment protocol will be carried out three times per week for 8 weeks
  Interventions: Other: Self-sinus massage technique

INTERVENTIONS:
Device: pulsed electromagnetic therapy — We will use the ASTAR Physio MG 827, a generator and 75 cm solenoid couch, in a pulsed electromagnetic field group. Participants will be placed comfortably in the solenoid, and the device will be turned on and programmed for 20 guesses for 10 minutes, 7 Hz, three times per week for 8 weeks.
  Arms: pulsed electromagnetic therapy
Device: Photobiostimulation — The therapy will be performed using an ASTAR PhysioGo -As low level laser therapy device with a wavelength of 830 nm, 30 mW power output, and 1 J energy dose. Patients will be supine and wear laser safety goggles. The laser will be applied to six locations over the maxillary or frontal sinuses, administered in a continuous manner for 33 seconds per spot, totaling 198 seconds and 6 J per session
  Arms: Photobiostimulation
Other: Self-sinus massage technique — Participants are instructed to perform self-massage to their frontal and maxillary sinuses at home twice daily, in the morning and evening. For the frontal sinus, place the fingers above the eyebrows on either side of the forehead, and gently circular outward massage for three sets of 30 seconds, repeated twice a day.
  Arms: Self-sinus massage technique

SUMMARY:
This study was done to find out the effect of photobiostimulation and pulsed electromagnetic field in patients with chronic rhinosinusitis on:

* Quality of life.
* Pulmonary function.
* Mean platelet volume.
* headache .
* total nasal symptoms.

DETAILED DESCRIPTION:
Chronic rhinosinusitis is a severe disease that significantly impacts a patient's quality of life, leading to significant economic impacts on healthcare resources and absenteeism. Symptoms interfere with daily activities and can lead to medication resistance. Treatment options like steroids, oral antibiotics, and sinus surgery are less effective, and disease recurrence remains high even after surgery. Alternative therapies like low-level laser therapy and pulsed electromagnetic filed have shown promise in improving symptoms and potentially making low-level laser therapy a non-invasive treatment for Chronic rhinosinusitis

ELIGIBILITY:
Inclusion Criteria:

1. Participants suffering from mild to moderate symptoms (baseline Total nasal symptoms score ≤ 9).
2. Subjects age range from 20 to 40 years old.
3. Patients of both sexes.
4. proven positive allergy test (skin prick test or multiple allergen simultaneous test) to any of the common perennial allergens such as dust mites, molds, insects, and animal dander within the last 12 months

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Patients with a definite deviated nasal septum, or history of operation within the last 6 months.
* Hypertension, diabetes mellitus, malignancy, active pulmonary tuberculosis, active respiratory disease like asthma, or other systemic diseases.
* Long-term use of corticosteroids or immunosuppressive agents.
* Participation in another clinical study within 30 days.
* Hyperthyroidism
* Patients who had used antihistamines within 1 week, topical corticosteroids within 2 weeks, systemic corticosteroids within 4 weeks, anticholinergic drugs within 3 days, antileukotriene drugs within 1 week, decongestants within 3 days, tricyclic antidepressants or phenothiazines within 2 weeks, nonsteroidal analgesics within 2 weeks, and other drugs that the researchers believed were inappropriate.
* Patients with Tattoos, moles and dark skin

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
assessment of change of quality of life | at baseline and after 8 weeks
  The Sinonasal Outcome Test-22 questionnaire is a commonly used tool in clinical practice to assess patients' quality of life with chronic respiratory syndrome. It consists of 22 chronic respiratory syndrome-related items, ranging from 0 to 5, and categorizes them into physical symptoms (items 1-12) and health and quality of life (items 13-22), covering sleep function and psychological difficulties. It is easy to understand and complete.

SECONDARY OUTCOMES:
assessment of change of pulmonary functions | at baseline and after 8 weeks
  The Global Initiative for Chronic Obstructive Lung Disease 2010 guidelines outline a procedure for a spirometer. The patient is instructed to breathe in until their lungs feel full, then hold their breath tightly around the mouthpiece. The operator blasts the air out forcefully, encouraging the patient to continue. The procedure is repeated twice until three repeatable blows are obtained, with the best two readings within 150 mL or 5% of each other.
assessment of change of Mean platelet volume | at baseline and after 8 weeks
  Venous blood samples will be drawn to assess and calculate the average volume of individual platelets
assessment of change of white blood cells count | at baseline and after 8 weeks
  Venous blood samples will be drawn to assess and calculate the white blood cells count
assessment of change of headache pain severity | at baseline and after 8 weeks
  It will be used to evaluate headache pain severity using a standard horizontal scale as mild (1-3 on a visual analogue scale), moderate (4-6 on a visual analogue scale), severe (7-9 on a visual analogue scale) and very severe (10 on a visual analogue scale)
assessment of change of total nasal symptoms | at baseline and after 8 weeks
  It is the sum of scores for nasal congestion, sneezing, nasal itching, and rhinorrhea at each time point, using a four-point scale (0-3). A score of 0 indicates no symptoms, a score of 1 indicates mild symptoms that are easily tolerated, a score of 2 indicates awareness of bothersome but tolerable symptoms, and a score of 3 indicates severe symptoms that interfere with daily activities. The total nasal symptoms scale is calculated by combining the scores for each symptom to a total of 12

CONTACTS AND LOCATIONS:
Locations (1):
- out-patient clinic, faculty of physical therapy, October University for Modern Sciences and Arts, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No